CLINICAL TRIAL: NCT01742221
Title: A Phase 1b, Single-Dose, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HemaMax™ (rHuIL-12) in Healthy Subjects
Brief Title: Safety and Tolerability of HemaMax™ (rHuIL-12) as Radiation Countermeasure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neumedicines Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-002
Record Dates: First submitted 2012-08-06; First posted 2012-12-05 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Hematopoietic Syndrome Due to Acute Radiation Syndrome
Keywords: HemaMax, NM-IL-12, HSARS, Safety
MeSH Terms: interventions — Interleukin-12 Subunit p35

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HemaMax (Experimental): Single subcutaneous 12 microgram dose of HemaMax
  Interventions: Biological: HemaMax
- Placebo (Placebo Comparator): Single subcutaneous dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: HemaMax — single subcutaneous 12 microgram dose of HemaMax
  Other Names: rHuIL-12, NM-IL-12
  Arms: HemaMax
Drug: Placebo — single subcutaneous dose
  Arms: Placebo

SUMMARY:
This trial is designed to evaluate the safety, pharmacokinetics, and pharmacodynamics of HemaMax in healthy male and female volunteers.

DETAILED DESCRIPTION:
A randomized, placebo-controlled, double-blind study of HemaMax to evaluate the safety, tolerability, pharmacokinetics, immunogenicity and pharmacodynamics of a single 12 μg subcutaneous dose of HemaMax on 60 healthy subjects for 28 days after HemaMax administration.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects, who have signed the informed consent form must meet all of the following criteria

  1. 18 to 45 years of age
  2. Body mass index (BMI) > 19 and < 0 kg/m2
  3. Normal ECG, vital signs and laboratory test results
  4. Use of effective birth control method and abstinence from sex
  5. Negative pregnancy test and drug screen

Exclusion Criteria:

* Subjects with any of the following characteristics will be considered ineligible:

  1. History of clinically significant renal, hepatic pulmonary, cardiovascular, cerebrovascular, gastrointestinal, metabolic, hematological, endocrine, urological, immunological, neurologic or psychiatric disorders or connective tissue disease
  2. Positive for human immunodeficiency virus (HIV), Hepatitis B, or surface antigen (HBsAg) or Hepatitis C antibody, tuberculosis (TB)
  3. Current drug or alcohol addiction
  4. History of clinically significant allergy of any kind
  5. Prior use of IL-12 or HemaMax
  6. Use of any approved or investigational biologic agents or vaccinations of any kind in last 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of HemaMax in healthy subjects. | 3 months
  Number of subjects with adverse events as a measure of safety and tolerability

SECONDARY OUTCOMES:
To characterize the pharmacokinetics, pharmacodynamics and immunogenicity of HemaMax in healthy subjects | 3 months
  To evaluate PK parameters AUC, Cmax, Tmax, t ½, Vz/F, and CL/F for HemaMax. To evaluate biological response parameters following HemaMax.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Siebers, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gluzman-Poltorak Z, Vainstein V, Basile LA. Recombinant interleukin-12, but not granulocyte-colony stimulating factor, improves survival in lethally irradiated nonhuman primates in the absence of supportive care: evidence for the development of a frontline radiation medical countermeasure. Am J Hematol. 2014 Sep;89(9):868-73. doi: 10.1002/ajh.23770. Epub 2014 Jun 19. PMID 24852354
- [Background] Gluzman-Poltorak Z, Vainstein V, Basile LA. Association of Hematological Nadirs and Survival in a Nonhuman Primate Model of Hematopoietic Syndrome of Acute Radiation Syndrome. Radiat Res. 2015 Aug;184(2):226-30. doi: 10.1667/rr13962.1. Epub 2015 Jul 24. PMID 26207689
- [Background] Gluzman-Poltorak Z, Mendonca SR, Vainstein V, Kha H, Basile LA. Randomized comparison of single dose of recombinant human IL-12 versus placebo for restoration of hematopoiesis and improved survival in rhesus monkeys exposed to lethal radiation. J Hematol Oncol. 2014 Apr 6;7:31. doi: 10.1186/1756-8722-7-31. PMID 24708888
- [Background] Basile LA, Ellefson D, Gluzman-Poltorak Z, Junes-Gill K, Mar V, Mendonca S, Miller JD, Tom J, Trinh A, Gallaher TK. HemaMax, a recombinant human interleukin-12, is a potent mitigator of acute radiation injury in mice and non-human primates. PLoS One. 2012;7(2):e30434. doi: 10.1371/journal.pone.0030434. Epub 2012 Feb 24. PMID 22383962
- [Derived] Gokhale MS, Vainstein V, Tom J, Thomas S, Lawrence CE, Gluzman-Poltorak Z, Siebers N, Basile LA. Single low-dose rHuIL-12 safely triggers multilineage hematopoietic and immune-mediated effects. Exp Hematol Oncol. 2014 Apr 11;3(1):11. doi: 10.1186/2162-3619-3-11. PMID 24725395